CLINICAL TRIAL: NCT03661684
Title: Glucocorticoid Effects in Patients With DM Type 2
Brief Title: Effect of Short Course of Glucocorticoid in Patients With Diabetes Mellitus(DM) Type 2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Yannis Guerra, Endocrinology Attending, Cook County Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-035
Record Dates: First submitted 2017-06-01; First posted 2018-09-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Diabetes; Hyperglycemia Steroid-induced
Keywords: Diabetes; Glucocorticoids; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Two groups. Condition group and Control group, both receiving the investigated medication using the same protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prednisone in subjects with Diabetes (Experimental): Group of subjects with diabetes mellitus type 2 receiving prednisone 40 mg po q day for 3 days
  Interventions: Drug: Prednisone
- Prednisone in control subjects (Experimental): Group of subjects without diabetes mellitus type 2 receiving prednisone 40 mg po q day for 3 days
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — 40 mg po q day of Prednisone for 3 days
  Other Names: Deltasone, Prednicot, Rayos

SUMMARY:
Participants will receive prednisone 40 mg for 3 days. 75 g oral glucose tolerance test (OGTT), insulin and C-peptide will be measured on day 1 (before prednisone) and day 3 (after prednisone). Also capillary glucose values will be obtained during and after the period of prednisone intake.

DETAILED DESCRIPTION:
On their scheduled day, participants will be instructed to come to the clinic after an overnight fast of a minimum of 8 hours (subjects can drink water). The participants will be asked to refrain from drinking alcohol for a period of 24 hours before the study days and to not perform strenuous exercise for a period of 48 hours before the study days. The participants will be directed to avoid alcohol and strenuous exercise for the duration of the study.

On days 1 and 3 of the study period, participants will be checked into the clinic. A physical examination, including height, weight and waist circumference, and finger-stick glucose will be performed. A 75-g OGTT will be performed with venous samples for measurement of glucose, insulin and C-peptide levels obtained at 0, 30 and 60 minutes starting immediately after the ingestion of the 75 g glucose solution. After samples are collected on day 1, participants will be administered their first dose of steroid, prednisone 40 mg, and be given a packet of two additional doses for the rest of the study period. The investigators may only give 1 additional dose to them and have the participants take the last dose in clinic on day 3 two hours before the OGTT. Subjects will take prednisone 40 mg once daily for three days to be consumed around 8:00am on days 2 and 3. This dose was chosen as a typical high-dose glucocorticoid regimen. On the third day, the participants will again visit the clinic after an overnight fast of a minimum 8 hours and undergo a physical examination and OGTT just as on day 1.

Participants will be instructed to check pre-prandial (before breakfast, lunch and dinner), and bed time (around 10:00 pm) blood glucose (BG) levels and to record all values for a total of five days (three days while on prednisone and for two days after the second study visit). A member of the study staff will call each participant daily around 7:00 pm to obtain BG values. Compliance with the study protocol will be assessed at this time as well. Any subject not compliant with study medications will be excluded from the study.

ELIGIBILITY:
Experimental Group

Inclusion Criteria:

1. Males or non-pregnant females between the ages of 18-50 years being followed in the Diabetes Center.
2. Type 2 Diabetes for ≤ 1 year and only on metformin
3. BMI 24.0-35.0 kg/ m2
4. HBA1c ≤ 9.0%

Exclusion Criteria:

1. Patients on any other antidiabetes medication.
2. Patients with impaired renal function (estimated Glomerular Filtration Rate (GFR) less than 60 ml/min based on results from Cerner).
3. Patient who have received glucocorticoid therapy within six months of study.
4. Patients who do shift work.
5. Blood glucose level ≥ 250 mg/dl on finger-stick at clinic visit.
6. Signs or symptoms of infection.

Control Group

Inclusion Criteria:

1. Males or non-pregnant females between the ages of 18-50 years in good physical health as determined by medical history, physical examination, and screening blood tests
2. Normoglycemia defined by fasting plasma glucose < 5.6 mmol/L (or 100 mg/dL) and 2h glucose <7.8 mmol/L (or 140 mg/dL) after a 75 g OGTT
3. BMI: 22.0 - 28.0 kg/m2

Exclusion Criteria:

1. Presence of any disease or use of any medication
2. Patients with a first-degree relative with Type 2 Diabetes
3. Patients who smoke
4. Patients with history of steroid use in previous 6 months.
5. Patients who do shift work
6. Signs or symptoms of infection.
7. Patients with recent changes in weight or physical activity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
AUC for glucose during OGTT | Throughout the course of 3 days
  Comparison of the Area under the curve (AUC) of the OGTT for glucose values at 60 and 120 throughout the course of 3 days

SECONDARY OUTCOMES:
HOMA index | At day 1 and at day 3
  Comparison of Homeostatic model assessment (HOMA) index before and after receiving the prednisone dose (at day 1 and at day 3)
AUC for Insulin during OGTT | Throughout the course of 3 days
  Comparison of the Area under the curve of the OGTT for glucose values at 60 and 120 minutes throughout the course of 3 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donihi AC, Raval D, Saul M, Korytkowski MT, DeVita MA. Prevalence and predictors of corticosteroid-related hyperglycemia in hospitalized patients. Endocr Pract. 2006 Jul-Aug;12(4):358-62. doi: 10.4158/EP.12.4.358. PMID 16901792
- [Background] Hwang JL, Weiss RE. Steroid-induced diabetes: a clinical and molecular approach to understanding and treatment. Diabetes Metab Res Rev. 2014 Feb;30(2):96-102. doi: 10.1002/dmrr.2486. PMID 24123849
- [Background] van Raalte DH, Brands M, van der Zijl NJ, Muskiet MH, Pouwels PJ, Ackermans MT, Sauerwein HP, Serlie MJ, Diamant M. Low-dose glucocorticoid treatment affects multiple aspects of intermediary metabolism in healthy humans: a randomised controlled trial. Diabetologia. 2011 Aug;54(8):2103-12. doi: 10.1007/s00125-011-2174-9. Epub 2011 May 12. PMID 21562755
- [Derived] Shah M, Adel MM, Tahsin B, Guerra Y, Fogelfeld L. Effect of short-term prednisone on beta-cell function in subjects with type 2 diabetes mellitus and healthy subjects. PLoS One. 2020 May 5;15(5):e0231190. doi: 10.1371/journal.pone.0231190. eCollection 2020. PMID 32369480